CLINICAL TRIAL: NCT02556151
Title: Neuromodulation Therapy for Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: University of Manchester (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21DK104127-01 (NIH); 1R21DK104127-01 (NIH)
Record Dates: First submitted 2015-09-17; First posted 2015-09-22 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Hz (Active Comparator): Six sessions of weekly therapy with 1 Hz magnetic stimulations of the lumbar and sacral regions.
  Interventions: Procedure: Repetitive lumbosacral magnetic stimulation (rTLSMS)
- 5 Hz (Active Comparator): Six sessions of weekly therapy with 5 Hz magnetic stimulations of the lumbar and sacral regions.
  Interventions: Procedure: Repetitive lumbosacral magnetic stimulation (rTLSMS)
- 15 Hz (Active Comparator): Six sessions of weekly therapy with 15 Hz magnetic stimulations of the lumbar and sacral regions.
  Interventions: Procedure: Repetitive lumbosacral magnetic stimulation (rTLSMS)

INTERVENTIONS:
Procedure: Repetitive lumbosacral magnetic stimulation (rTLSMS) — Patients randomized to Six sessions of weekly therapy with either 1 HZ or 5 Hz or 15 Hz magnetic stimulations of the lumbar and sacral regions.
  Other Names: rTLSMS

SUMMARY:
Fecal Incontinence (FI) affects 8-15 % of the US population, predominantly women and elderly, and 45% of nursing home residents. It significantly impairs quality of life and poses a major health care burden. FI is characterized by significant neuromuscular dysfunction of the pelvic floor that includes bilateral lumbo-anorectal and sacro-anorectal neuropathy and sensori-motor dysfunction. This multifactorial etiology suggests that maladaptive neuroplastic changes in the neural innervation of lower gastrointestinal tract could play a significant role in the pathogenesis of FI. A critical barrier to progress in the treatment of FI is the lack of understanding of how treatments affect the core pathophysiological mechanisms of FI, and the absence of mechanistically based non-invasive therapies. Our goal is to address the problem of FI by developing therapies that modulate peripheral and central neuronal perturbations and thereby improve visceromotor control and sensori-motor dysfunctions, and to understand the neurobiologic basis of these treatments. Our central hypothesis is that a novel non-invasive treatment consisting of repetitive translumbar magnetic stimulation (rTLMS) and repetitive transsacral magnetic stimulation (rTSMS) will significantly improve FI by enhancing peripheral and central neural excitability and will provide a multidimensional therapeutic benefit- enhance anal muscle strength, improve stool perception and improve rectal capacity. Our approach is based on our preliminary studies which suggest that repetitive translumbar magnetic stimulation (rTLMS) and transsacral magnetic stimulation (rTSMS) improve anorectal pain and neuropathy and induce central neuroplastic changes.

Our objectives are to:

1. address the significant gap in our knowledge regarding the peripheral and central neuroenteric axis and how perturbations in the afferent and efferent neural signaling can affect FI;
2. develop a new treatment for FI with repetitive magnetic stimulation and determine the feasibility, safety and optimal frequency setting of rTLMS and rTSMS;
3. determine the mechanistic basis for this neuromodulation therapy;
4. identify if the locus for improvement lies in the afferent or efferent signaling or both.

DETAILED DESCRIPTION:
Our expected outcome include development of new treatment approaches for FI which are mechanistically based, effective, safe, low cost, less invasive, low risk and less dependent on patient compliance.

The impact of our project include a new non-invasive treatment modality for FI, a scientific basis for the development of this treatment and improved understanding of the peripheral and central neuroenteric axis in FI.

Aim 1: Test the hypothesis that neuromodulation therapy with combined repetitive translumbar magnetic stimulation (rTLMS) and transsacral magnetic stimulation (rTSMS) improves symptoms in FI patients. Investigators will evaluate the efficacy, safety and optimal frequency setting of rTLMS and rTSMS for FI by investigating whether 6 sessions of weekly therapy with 1 Hz or 5Hz or 15 Hz magnetic stimulations of the lumbar and sacral regions provides therapeutic response in FI patients. Investigators will randomize 48 patients with FI and assess symptoms and anorectal function. The primary outcome measure will be the reduction in number of episodes of FI. The secondary outcome measures will be i) bowel symptoms/severity (FISI, FICA), ii) quality-of-life (FI-QOL), iii) psychosocial function, iv) anal sphincter pressures, v) rectal sensation, vi) rectal compliance. A safety assessment will monitor adverse effects.

Aim 2: Test the hypothesis that repetitive translumbar magnetic stimulation (rTLMS) and transsacral magnetic stimulation (rTSMS) will improve FI symptoms and anorectal function through modulation of ascending and descending signaling pathways in the neuroenteric axis. Investigators will investigate the mechanistic basis for rTLMS/rTSMS therapy by examining the neuroenteric axis. Investigators will examine rectal and anal motor evoked potentials (MEPs) in 48 FI patients with transcranial, translumbar and transsacral magnetic stimulations (descending signaling), before and after 6 sessions of therapy with 1 Hz or 5 Hz or 15 Hz magnetic stimulations. Also, investigators will examine the cortical evoked potentials (CEP) after anal and rectal stimulation (ascending signaling). investigators will determine whether rTLMS and rTSMS therapy shortens latency and increases amplitude and area under curve (AUC) of anal and rectal MEPs and ano-cortical and recto-cortical CEPs when compared to baseline. Investigators will identify if the locus for improvement lies in the afferent signaling, efferent signaling or both and whether the neuroplastic changes are central or peripheral. The primary outcome measure for efferent signaling will be the latency of lumbo-anal and sacro-anal MEP responses and for afferent signaling will be the latency of ano-cortical CEP. Secondary outcome measures include anal and rectal electrical sensory thresholds, lumbo-rectal and sacro-rectal MEPs and recto-cortical CEPs and correlations of FI episodes and bowel symptoms with changes in latency and MEP measurements.

Participants will maintain a two week prospective fecal incontinence symptom diary. Baseline questionnaires will be administered. Patients demonstrating at least one episode of fecal incontinence per week, on average, will be eligible, pending all other eligibility criteria is met. Patients will come for brain-gut assessment (as above) as well as baseline anorectal manometry (if needed per protocol specifications). Patients will be randomized to one of the three hertz groups and have treatment one within one week of baseline assessments. A total of six weekly treatments (with a +7 day window allowed), will occur. After the six treatments, patients will have all baseline assessments repeated (brain-gut assessments, anorectal manometry and questionnaires).

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent episodes of FI for 6 months;
2. No mucosal disease (colonoscopy + biopsy); and
3. On a 2-week stool diary patients reported at least one episode of solid or liquid FI/week.

Exclusion Criteria: Patients with

1. severe diarrhea (>6 liquid stools/day, Bristol scale >6);
2. on opioids, tricyclics (except on stable doses > 3months);
3. active depression;
4. comorbid illnesses, severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy;
5. neurologic diseases (e.g. head injury, epilepsy, multiple sclerosis, strokes, spinal cord injury);
6. impaired cognizance (mini mental score of < 15/25) and/or legally blind;
7. metal implants, pacemakers;
8. previous pelvic surgery, bladder repair, radical hysterectomy;
9. ulcerative and Crohn's colitis;
10. rectal prolapse, anal fissure, anal surgery or inflamed hemorrhoids;
11. pregnant women
12. nursing mothers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The reduction in number of episodes of Fecal Incontinence | 12 weeks
  The primary outcome measure will be the reduction in number of episodes of Fecal incontinence from baseline to post treatment.

SECONDARY OUTCOMES:
Bowel symptoms | 12 weeks
  Changes from baseline in reporting of bowel symptoms/severity (FICA)
Fecal incontinence Quality of life | 12 weeks
  Changes from baseline in quality-of-life domains (FI-QOL)
Psychosocial function | 12 weeks
  Changes from baseline in psychological report symptoms (Rome Psychosocial Assessment)
Anal and rectal sensations | 12 weeks
  Changes from baseline on anorectal manometry

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, MD, PhD, Principal Investigator — Augusta University
Locations (2):
- Augusta University, Augusta, Georgia, United States
- University of Manchester, Manchester, United Kingdom